CLINICAL TRIAL: NCT03435276
Title: A Phase 1, Randomized, Placebo-controlled Study to Assess the Safety, Tolerability and Pharmacokinetics of AZD9977 Following Multiple-Ascending Dose Administration in Healthy Volunteers
Brief Title: Multiple-ascending Dose Study to Assess the Safety, Tolerability and Pharmacokinetics of AZD9977 in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D6401C00001
Record Dates: First submitted 2018-01-25; First posted 2018-02-19 (Actual); Last update posted 2018-06-21 (Actual); Status verified 2018-06

CONDITIONS: Healthy Volunteers
Keywords: Heart failure.; Oral selective mineralocorticoid receptor modulator.; Heart failure with preserved ejection fraction (HFpEF).
MeSH Terms: conditions — Heart Failure | interventions — AZD9977

STUDY DESIGN:
Who Masked: Participant
Masking Description: This study is single-blind (in which the study center staff have to remain blinded during the clinical conduct of a given cohort) with regard to treatment (AZD9977 or placebo) at each dose level. In the event of a medical emergency when management of a subject's condition requires knowledge of the trial medication, the treatment received may be revealed by personnel authorized by the PI. Reasons for breaking a code will be clearly explained and justified in ClinBase. The date on which the code was broken together with the identity of the person responsible will also be documented.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): Randomized subjects will receive AZD9977 50 mg or placebo oral suspension single dose on Day 1 and Day 8; twice daily dose Day 2 to Day 7
  Interventions: Drug: AZD9977; Other: Placebo
- Cohort 2 (Experimental): Randomized subjects will receive AZD9977 150 mg or placebo oral suspension single dose on Day 1 and Day 8; twice daily dose on Day 2 to Day 7
  Interventions: Drug: AZD9977; Other: Placebo
- Cohort 3 (Experimental): Randomized subjects will receive AZD9977 300 mg or placebo oral suspension single dose on Day 1 and Day 8; twice daily dose on Day 2 to Day 7
  Interventions: Drug: AZD9977; Other: Placebo

INTERVENTIONS:
Drug: AZD9977 — Randomized subjects will receive AZD9977 oral suspension at a dose of 50 mg in Cohort 1, 150 mg in Cohort 2 and 300 mg in Cohort 3
Other: Placebo — Randomized subjects will receive orally AZD9977 matched placebo in Cohorts 1, 2 and 3

SUMMARY:
This is a randomized, single-blind, placebo-controlled study conducted on healthy male subjects at a single study center to assess the safety, tolerability and the pharmacokinetics of AZD9977 following multiple-ascending oral doses at steady state

DETAILED DESCRIPTION:
This is a phase 1, randomized, single-blind, placebo-controlled, single center, multiple-ascending dose sequential-group design study conducted on 45 healthy male subjects to investigate the safety, tolerability, pharmacokinetics (PK) of AZD9977, time to reach steady state, the degree of accumulation and the time dependency of the PK. The study consists of three visits:

* A screening period (maximum 28 days)
* A treatment period (subjects will be resident from 2 days before first dose of investigation medicinal product (IMP) (Day -2) until at least 36 after last dose of IMP and will be discharged on Day 9) and
* A follow-up visit within 5 to 7 days after last dose of IMP. This study consists of 3 Cohorts (9 subjects each). Based on the safety review committee (SRC) requirement, 2 additional cohorts may be added either to repeat a dose level or additional dose steps, if required. In each cohort, subjects will be randomized to receive AZD9977 (6 subjects) and placebo (3 subjects) oral suspension twice daily. The dose of AZD9977 in Cohort 1 will be 50 mg as starting dose and in Cohort 2 and 3 at provisional dose 150 mg and 300 mg, respectively. Each subject will receive a total of 14 oral doses of AZD9977 or placebo. Each subject will receive a single dose of IMP in the morning of Day 1 and Day 8 and twice daily doses on Day 2 to Day 7.

On Day 1 and Day 8, subjects will be fasted for 10 hours before dosing until 4 hours after dosing when lunch will be served. On Day 2 to Day 6, subjects will be fasted for 10 hours before dosing until 1 hour after dosing when breakfast will be served. On Day 7, subjects will be fasted for 10 hours before dosing and until after the completion of the oral glucose tolerance test (OGTT) when breakfast will be served. For the evening dose of IMP (Days 2 to Day 7), subjects will be fasted for 2 hours before dosing until 1 hour after dosing. On all days, subjects will be allowed to drink freely until 1 hour before dosing to prevent dehydration before each morning and evening dose and water consumption could be resumed 1 hour after dosing.

Dosing for each ascending dose cohort will proceed with 2 subjects in a sentinel cohort, such that 1 subject will be randomized to receive placebo and 1 subject will be randomized to receive AZD9977. The safety data from the sentinel subjects up to 72 hours post first dose will be reviewed by the principal investigator (PI) before the remaining subjects in the cohort are dosed. Following review of data from the study, the SRC may decide to adjust the length of the stay at the study site and the timing and number of assessments and/or blood samples for subsequent cohorts. The time window between the single dose and start of repeated dosing may also be adjusted. The duration of the study is approximately 6 weeks

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated, written informed consent before any study specific procedures.
2. Healthy male subject aged 18 to 50 years (inclusive) with suitable veins for cannulation or repeated venipuncture.
3. Have a body mass index (BMI) between 18 and 30 kg/m2(inclusive) and weigh at least 50 kg and no more than 100 kg (inclusive).
4. Provision of signed, written and dated informed consent for optional genetic and/or biomarker research. If a subject declines to participate in the genetic components of the study, there will be no penalty or loss of benefit to the subject. The subject will not be excluded from other aspects of the study.

Exclusion Criteria:

1. History of any clinically important disease/disorder which, in the opinion of the Investigator, may either put the subject at risk because of participation in the study/influence the results/subject's ability to participate in the study.
2. History/presence of gastrointestinal, hepatic/renal disease/any other condition known to interfere with absorption, distribution, metabolism/excretion of drugs.
3. Any clinically important illness, medical/surgical procedure or trauma within 4 weeks of the 1st administration of the IMP.
4. Any clinically important abnormalities in clinical chemistry, hematology or urinalysis results at the Screening Visit and/or admission, as judged by the Investigator and specified below: Serum potassium > 5.0 mmol/L; Hemoglobin A1c (HbA1c) > 5.7%.
5. Any positive result on screening for serum hepatitis B surface antigen, hepatitis C antibody & human immunodeficiency virus (HIV).
6. Abnormal vital signs, after 10 minutes supine rest at the Screening Visit and/or admission, defined as any of the following: Systolic BP < 90 mmHg or > 140 mmHg; Diastolic BP < 50 mmHg or > 90 mmHg; Heart rate < 45 or > 85 beats per minute (bpm).
7. Any clinically important abnormalities in rhythm, conduction or morphology of the resting ECG and any clinically important abnormalities in the 12-lead ECG as judged by the Investigator that may interfere with the interpretation of QTc interval changes, including abnormal ST-T-wave morphology, particularly in the CSP defined primary lead or LV hypertrophy at the Screening Visit or/and admission.

   * Prolonged QT interval corrected for HR by Fridericia's formula (QTcF) > 450 ms or shortened QTcF < 340 ms or family history of long QT syndrome.
   * PR (PQ) interval shortening < 120 ms (PR > 110 ms but < 120 ms is acceptable if there is no evidence of ventricular preexcitation).
   * PR (PQ) interval prolongation (> 240 ms intermittent second (Wenckebach block while asleep is not exclusive) or 3rd degree atrioventricular (AV) block, or AV dissociation.
   * Persistent/intermittent complete bundle branch block (BBB), incomplete bundle branch block (IBBB), or intraventricular conduction delay (IVCD) with QRS > 110 ms. Subjects with QRS > 110 ms but < 115 ms are acceptable if there is no evidence of ventricular hypertrophy or pre-excitation.
8. Known or suspected history of drug abuse in the last 12 months before the Screening Visit as judged by the Investigator.
9. Current smokers/those who have smoked/used nicotine products (including e-cigarettes) within last 3 months before the Screening Visit.
10. History of alcohol abuse in the last 12 months before the Screening Visit/current excessive intake of alcohol as judged by the Investigator.
11. Positive screen for drugs of abuse, alcohol/cotinine (nicotine) at the Screening Visit/admission.
12. History of severe allergy/hypersensitivity or ongoing clinically important allergy/hypersensitivity, as judged by the Investigator or history of hypersensitivity to drugs with a similar chemical structure or class to AZD9977.
13. Excessive intake of caffeine-containing drinks/food (e.g., coffee, tea, chocolate,) as judged by the Investigator.
14. Use of drugs with enzyme inducing properties like St John's Wort within 3 weeks before the 1st administration of the IMP.
15. Use of any prescribed/non-prescribed medication including antacids, analgesics (other than paracetamol/acetaminophen), herbal remedies, megadose vitamins (intake of 20 to 600 times the recommended daily dose) and minerals during the 2 weeks before the first administration of the IMP or longer if the medication has a long half-life.
16. Plasma donation within 1 month of the Screening Visit or any blood donation/blood loss > 500 mL during the 3 months before the Screening Visit.
17. Has received another new chemical/non-chemical entity (a compound which has not been approved for marketing) within 3 months of the first administration of IMP in this study. The exclusion period 3 months after the final dose/1 month after the last visit whichever is the longest.
18. Subjects who have previously received AZD9977.
19. Involvement of any Astra Zeneca or study site employee or their close relatives.
20. Judgment by the Investigator that the subject should not participate in the study if they have any ongoing/recent (during the Screening period) minor medical complaints that may interfere with the interpretation of study data or are considered unlikely to comply with study procedures, restrictions and requirements.
21. Subjects who cannot communicate reliably with the Investigator.
22. Vulnerable subjects (kept in detention, protected adults under guardianship, trusteeship or committed to an institution by governmental or juridical order).
23. Previous bone marrow transplant.
24. Non-leukocyte depleted whole blood transfusion within 120 days of the date of the genetic sample collection.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2018-02-27 (Actual); Primary Completion 2018-06-13 (Actual); Study Completion 2018-06-13 (Actual)

PRIMARY OUTCOMES:
Number of subjects with adverse events (AEs) due to AZD9977 | From baseline up to follow-up (5 to 7 days post last dose)
  To assess AEs as variable of safety and tolerability after administration of multiple dose of AZD9977 oral suspension. AEs will be collected from the start of screening throughout the treatment period up to and including the follow-up visit. Serious AEs will be recorded from the time of informed consent.
Systolic blood pressure [SBP] | From baseline up to follow-up (5 to 7 days post last dose)
  To measure SBP as variable of safety and tolerability after administration of multiple dose of AZD9977 oral suspension. SBP will be collected after the subject has rested in the supine position for at least 10 minutes.
Diastolic blood pressure [DBP] | From baseline up to follow-up (5 to 7 days post last dose)
  To measure DBP as variable of safety and tolerability after administration of multiple dose of AZD9977 oral suspension. DBP will be collected after the subject has rested in the supine position for at least 10 minutes.
Pulse rate | From baseline up to follow-up (5 to 7 days post last dose)
  To measure pulse as variable of safety and tolerability after administration of multiple dose of AZD9977 oral suspension. Pulse rate will be collected after the subject has rested in the supine position for at least 10 minutes.
Laboratory assessments of urine volume | From baseline up to follow-up (5 to 7 days post last dose)
  To assess the urine volume as variable of safety and tolerability after administration of multiple dose of AZD9977 oral suspension.
Number of participants with abnormal findings in Twelve-lead (12-Lead) electrocardiograms (ECGs) (safety ECGs and 12-lead continuous digital ECG [dECG]) | From baseline up to follow-up (5 to 7 days post last dose)
  To assess any clinically significant abnormalities on cardiac electrophysiological parameters as variables of safety and tolerability after administration of multiple dose of AZD9977 oral suspension. 12-lead safety ECG and dECG will be obtained after the participant rested in the supine position for at least 10 minutes. Safety ECG will be collected at the end of each dECG recording. Various dECG variables like time between 2 consecutive R waves on ECG (RR), ECG interval measured form onset of P wave to the onset of QRS complex (PR), ECG interval measured from onset of QRS complex to the J point (QRS) and ECG interval measured form onset of QRS complex to the end of the T wave (QT intervals) will be reported. Derived parameters like QT interval corrected for heart rate using Fridericia's formula (QTcF), heart rate (HR) and others, as applicable are also calculated.
Number of participants with abnormal cardiac telemetry | From baseline up to follow-up (5 to 7 days post last dose)
  To assess any clinically significant abnormalities in the cardiovascular system functioning as variables of safety and tolerability after administration of multiple dose of AZD9977 oral suspension. A 2-lead real-time telemetry ECG will be used to assess the heart rate.
Number of participants with abnormal physical examination findings | From baseline up to follow-up (5 to 7 days post last dose)
  To assess any clinically significant abnormal physical examination findings as a variable of safety and tolerability after administration of multiple dose of AZD9977 oral suspension. Brief physical examination includes assessment of the general appearance, skin, cardiovascular system, respiratory and abdomen. Full physical examination includes assessment of the general appearance, skin, cardiovascular, respiratory, abdomen, head and neck (including ears, eyes, nose and throat), lymph nodes, thyroid, musculoskeletal and neurological systems.
Laboratory assessments: Hematology - Differential count | From baseline up to follow-up (5 to 7 days post last dose)
  To assess the differential white blood cell count (absolute count of basophils, eosinophils, lymphocytes, monocyets and neutrophils) as variables of safety and tolerability after administration of multiple dose of AZD9977 oral suspension.
Laboratory assessments: Hematology - Hematocrit (HCT) and Reticulocyte absolute count | From baseline up to follow-up (5 to 7 days post last dose)
  To assess the HCT (red blood cells [RBC]) and reticulocyte absolute count (immature RBCs) as variables of safety and tolerability after administration of multiple dose of AZD9977 oral suspension.
Laboratory assessments: Hematology - Hemoglobin (Hb) | From baseline up to follow-up (5 to 7 days post last dose)
  To assess the Hb as variables of safety and tolerability after administration of multiple dose of AZD9977 oral suspension.
Laboratory assessments: Hematology - Mean corpuscular hemoglobin (MCH) | From baseline up to follow-up (5 to 7 days post last dose)
  To assess the MCH as variables of safety and tolerability after administration of multiple dose of AZD9977 oral suspension.
Laboratory assessments: Hematology - Mean corpuscular hemoglobin concentration (MCHC) | From baseline up to follow-up (5 to 7 days post last dose)
  To assess the MCHC as variables of safety and tolerability after administration of multiple dose of AZD9977 oral suspension.
Laboratory assessments: Hematology - Mean corpuscular volume (MCV) | From baseline up to follow-up (5 to 7 days post last dose)
  To assess the MCV as variables of safety and tolerability after administration of multiple dose of AZD9977 oral suspension.
Laboratory assessments: Hematology - Platelets | From baseline up to follow-up (5 to 7 days post last dose)
  To assess platelets count as variables of safety and tolerability after administration of multiple dose of AZD9977 oral suspension.
Laboratory assessments: Hematology - Blood cells count | From baseline up to follow-up (5 to 7 days post last dose)
  To assess RBC and white blood cells (WBC) count as variables of safety and tolerability after administration of multiple dose of AZD9977 oral suspension.
Laboratory assessments: Serum Clinical chemistry - Albumin | From baseline up to follow-up (5 to 7 days post last dose)
  To assess the serum albumin level as variables of safety and tolerability after administration of multiple dose of AZD9977 oral suspension.
Laboratory assessments: Serum Clinical chemistry - C reactive protein (CRP) | From baseline up to follow-up (5 to 7 days post last dose)
  To assess the serum CRP level as variables of safety and tolerability after administration of multiple dose of AZD9977 oral suspension.
Laboratory assessments: Serum Clinical chemistry - Creatine kinase (CK) | From baseline up to follow-up (5 to 7 days post last dose)
  To assess the serum CK level as variables of safety and tolerability after administration of multiple dose of AZD9977 oral suspension.
Laboratory assessments: Serum Clinical chemistry - Creatinine | From baseline up to follow-up (5 to 7 days post last dose)
  To assess the serum creatinine level as variables of safety and tolerability after administration of multiple dose of AZD9977 oral suspension.
Laboratory assessments: Serum Clinical chemistry - Glucose (fasting) | From baseline up to follow-up (5 to 7 days post last dose)
  To assess the serum fasting glucose level as variables of safety and tolerability after administration of multiple dose of AZD9977 oral suspension.
Laboratory assessments: Serum Clinical chemistry - Calcium, potassium, phosphate and sodium | From baseline up to follow-up (5 to 7 days post last dose)
  To assess the serum calcium, potassium, phosphate and sodium level as variables of safety and tolerability after administration of multiple dose of AZD9977 oral suspension.
Laboratory assessments: Serum Clinical chemistry - Urea and Uric acid | From baseline up to follow-up (5 to 7 days post last dose)
  To assess the serum urea and uric acid level as variables of safety and tolerability after administration of multiple dose of AZD9977 oral suspension.
Laboratory assessments: Serum Clinical chemistry - Liver enzymes | From baseline up to follow-up (5 to 7 days post last dose)
  To assess the serum Alanine aminotransferase (ALT), Alkaline phosphatase (ALP), Aspartate aminotransferase (AST) and Gamma glutamyl transpeptidase (GGT) level as variables of safety and tolerability after administration of multiple dose of AZD9977 oral suspension.
Laboratory assessments: Serum Clinical chemistry - Bilirubin | From baseline up to follow-up (5 to 7 days post last dose)
  To assess the serum bilirubin (total and unconjugated) level as variables of safety and tolerability after administration of multiple dose of AZD9977 oral suspension.
Laboratory assessments: Serum Clinical chemistry - Steroid | From baseline up to follow-up (5 to 7 days post last dose)
  To assess the serum cholesterol and triglycerides level as variables of safety and tolerability after administration of multiple dose of AZD9977 oral suspension.
Laboratory assessments: Serum Clinical chemistry - Luteinizing hormone (LH) | From baseline up to follow-up (5 to 7 days post last dose)
  To assess the serum LF level as variables of safety and tolerability after administration of multiple dose of AZD9977 oral suspension.
Laboratory assessments: Serum Clinical chemistry - Sex hormone binding globulin (SHBG) | From baseline up to follow-up (5 to 7 days post last dose)
  To assess the serum SHBG level as variables of safety and tolerability after administration of multiple dose of AZD9977 oral suspension.
Laboratory assessments: Serum Clinical chemistry - Testosterone | From baseline up to follow-up (5 to 7 days post last dose)
  To assess the serum testosterone level as variables of safety and tolerability after administration of multiple dose of AZD9977 oral suspension.
Laboratory assessments: Serum Clinical chemistry - Aldosterone | From baseline up to follow-up (5 to 7 days post last dose)
  To assess the serum aldosterone level as variables of safety and tolerability after administration of multiple dose of AZD9977 oral suspension.
Laboratory assessments: Serum Clinical chemistry - Hemoglobin A1c (HbA1c) | From baseline up to follow-up (5 to 7 days post last dose)
  To assess the serum HbA1c level as variables of safety and tolerability after administration of multiple dose of AZD9977 oral suspension.
Laboratory assessments: Serum Clinical chemistry - High-sensitivity troponin T | From baseline up to follow-up (5 to 7 days post last dose)
  To assess the serum high-sensitivity troponin T level as variables of safety and tolerability after administration of multiple dose of AZD9977 oral suspension.
Laboratory assessments: Serum Clinical chemistry - N-terminal pro-brain natriuretic peptide (NT-proBNP) | From baseline up to follow-up (5 to 7 days post last dose)
  To assess the serum NT-proBNP level as variables of safety and tolerability after administration of multiple dose of AZD9977 oral suspension.
Laboratory assessments: Serum Clinical chemistry - Follicle-stimulating hormone (FSH) | From baseline up to follow-up (5 to 7 days post last dose)
  To assess the serum FSH level as variables of safety and tolerability after administration of multiple dose of AZD9977 oral suspension.
Laboratory assessments: Clinical Urinalysis - Protein | From baseline up to follow-up (5 to 7 days post last dose)
  To assess the urine protein level as variables of safety and tolerability after administration of multiple dose of AZD9977 oral suspension. If urinalysis is positive for protein, a microscopy test will be performed to assess RBC, WBC, casts [cellular, granular, hyaline]).
Laboratory assessments: Clinical Urinalysis - Blood | From baseline up to follow-up (5 to 7 days post last dose)
  To assess the urine blood level as variables of safety and tolerability after administration of multiple dose of AZD9977 oral suspension. If urinalysis is positive for blood, a microscopy test will be performed to assess RBC, WBC, casts [cellular, granular, hyaline]).
Laboratory assessments: Clinical Urinalysis - Glucose | From baseline up to follow-up (5 to 7 days post last dose)
  To assess the urine glucose level as variables of safety and tolerability after administration of multiple dose of AZD9977 oral suspension.
Laboratory assessments: Clinical Urinalysis - Uric acid | From baseline up to follow-up (5 to 7 days post last dose)
  To assess the urine uric acid level as variables of safety and tolerability after administration of multiple dose of AZD9977 oral suspension.
Laboratory assessments: Clinical Urinalysis - Creatinine | From baseline up to follow-up (5 to 7 days post last dose)
  To assess the urine creatinine level as variables of safety and tolerability after administration of multiple dose of AZD9977 oral suspension.
Laboratory assessments: Urinalysis - Urinary Electrolytes | From baseline up to follow-up (5 to 7 days post last dose)
  To assess the urine electrolytes level (calcium, chloride, potassium and sodium) as variables of safety and tolerability after administration of multiple dose of AZD9977 oral suspension.

SECONDARY OUTCOMES:
Plasma PK parameter: Observed maximum plasma concentration (Cmax) | Treatment period:Day 1 and Day 8 (Pre-dose & 20 min, 40 min, 1, 2, 4, 6, 8, 10, 12, 16, & 20 hours post-dose)
  To assess Cmax after administration of multiple dose of AZD9977 oral suspension.
Plasma PK parameter: Time to reach maximum concentration (tmax) | Treatment period:Day 1 and Day 8 (Pre-dose & 20 min, 40 min, 1, 2, 4, 6, 8, 10, 12, 16, & 20 hours post-dose)
  To assess tmax after administration of multiple dose of AZD9977 oral suspension.
Plasma PK parameter: Terminal half-life (t1/2λz) | Treatment period:Day 1 and Day 8 (Pre-dose & 20 min, 40 min, 1, 2, 4, 6, 8, 10, 12, 16, & 20 hours post-dose)
  To assess t1/2λz after administration of multiple dose of AZD9977 oral suspension; estimated as (ln2)/λz
Plasma PK parameter: Terminal rate constant (λz) | Treatment period:Day 1 and Day 8 (Pre-dose & 20 min, 40 min, 1, 2, 4, 6, 8, 10, 12, 16, & 20 hours post-dose)
  To assess λz after administration of multiple dose of AZD9977 oral suspension; estimated by log-linear least squares regression of the terminal part of the concentration-time curve
Plasma PK parameter: Area under the plasma concentration-time curve in the dosing interval (AUCτ) | Treatment period:Day 1 and Day 8 (Pre-dose & 20 min, 40 min, 1, 2, 4, 6, 8, 10, 12, 16, & 20 hours post-dose)
  To assess AUCτ after administration of multiple dose of AZD9977 oral suspension.
Plasma PK parameter: Area under the plasma concentration-time curve from time zero to the time of the last measurable concentration (AUClast) | Treatment period:Day 1and Day 8 (Pre-dose & 20 min, 40 min, 1, 2, 4, 6, 8, 10, 12, 16, & 20 hours post-dose)
  To assess AUClast after administration of multiple dose of AZD9977 oral suspension.
Plasma PK parameter: Apparent volume of distribution for parent drug at terminal phase (Vz/F) | Treatment period:Day 1 and Day 8 (Pre-dose & 20 min, 40 min, 1, 2, 4, 6, 8, 10, 12, 16, & 20 hours post-dose)
  To assess Vz/F after administration of multiple dose of AZD9977 oral suspension, estimated by dividing the apparent
Plasma PK parameter: Apparent clearance for parent drug (CL/F) | Treatment period:Day 1 and Day 8 (Pre-dose & 20 min, 40 min, 1, 2, 4, 6, 8, 10, 12, 16, & 20 hours post-dose)
  To assess CL/F after administration of multiple dose of AZD9977 oral suspension, estimated as dose divided by AUC
Plasma PK parameter: Dose normalized AUCτ (AUCτ/D) | Treatment period:Day 1 and Day 8 (Pre-dose & 20 min, 40 min, 1, 2, 4, 6, 8, 10, 12, 16, & 20 hours post-dose)
  To assess AUCτ/D after administration of multiple dose of AZD9977 oral suspension, estimated by dividing AUCτ by the dose administered
Plasma PK parameter: Dose normalized Cmax (Cmax/D) | Treatment period:Day 1 and Day 8 (Pre-dose & 20 min, 40 min, 1, 2, 4, 6, 8, 10, 12, 16, & 20 hours post-dose)
  To assess Cmax/D after administration of multiple dose of AZD9977 oral suspension, estimated by dividing Cmax by the dose administered
Plasma PK parameter: Mean Residence Time (MRT) | Treatment period:Day 1 and Day 8 (Pre-dose & 20 min, 40 min, 1, 2, 4, 6, 8, 10, 12, 16, & 20 hours post-dose)
  To assess MRT after administration of multiple dose of AZD9977 oral suspension.
Plasma PK parameter: Area under the concentration-time curve from time zero extrapolated to infinity (AUC) | Treatment period:Day 1 (Pre-dose & 20 min, 40 min, 1, 2, 4, 6, 8, 10, 12, 16, & 20 hours post-dose)
  To assess AUC after administration of multiple dose of AZD9977 oral suspension. AUC is estimated by AUClast+ Clast/λz where Clast is the last observed quantifiable concentration
Plasma PK parameter: Dose normalized AUC (AUC/D) | Treatment period:Day 1 (Pre-dose & 20 min, 40 min, 1, 2, 4, 6, 8, 10, 12, 16, & 20 hours post-dose)
  To assess AUC/D after administration of multiple dose of AZD9977 oral suspension. AUC is estimated by dividing AUC by the dose administered.
Plasma PK parameter: Dose normalized AUClast (AUClast/D) | Treatment period:Day 1 (Pre-dose & 20 min, 40 min, 1, 2, 4, 6, 8, 10, 12, 16, & 20 hours post-dose)
  To assess AUClast/D after administration of multiple dose of AZD9977 oral suspension; estimated by dividing AUClast by the dose administered.
Plasma PK parameter: Observed concentration at the end of the dosing interval (Cmin) | Treatment period: Day 8 (Pre-dose & 20 min, 40 min, 1, 2, 4, 6, 8, 10, 12, 16, & 20 hours post-dose)
  To assess Cmin after administration of multiple dose of AZD9977 oral suspension.
Plasma PK parameter: Accumulation ratio for AUCτ (Rac AUCτ) | Treatment period: Day 8 (Pre-dose & 20 min, 40 min, 1, 2, 4, 6, 8, 10, 12, 16, & 20 hours post-dose)
  To assess Rac AUCτ after administration of multiple dose of AZD9977 oral suspension; estimated by dividing AUCτ from the last dosing day by AUCτ on Day 1
Plasma PK parameter: Accumulation ratio for AUCτ (Rac Cmax) | Treatment period: Day 8 (Pre-dose & 20 min, 40 min, 1, 2, 4, 6, 8, 10, 12, 16, & 20 hours post-dose)
  To assess Rac Cmax after administration of multiple dose of AZD9977 oral suspension; estimated by dividing maximum (peak) steady-state plasma drug concentration (Css,max) from the last dosing day by Cmax on Day 1
Plasma PK parameter: Temporal change (TCP) | Treatment period: Day 8 (Pre-dose & 20 min, 40 min, 1, 2, 4, 6, 8, 10, 12, 16, & 20 hours post-dose)
  To assess TCP after administration of multiple dose of AZD9977 oral suspension; estimated by dividing AUCτ from the last dosing day by AUC on Day 1
Urine PK parameter: Renal clearance (CLR) | Treatment period: Day 8 (Pre-dose and 0-4, 4-8 and 8-12 hours post-dose)
  To assess CLR after administration of multiple dose of AZD9977 oral suspension; estimated by dividing amount of analyte excreted into urine (Ae[0-t]) by AUC(0-t) where the time interval for both parameters are the same
Urine PK parameter: Amount of analyte excreted into the urine from time t1 to t2 (Ae[t1-t2]) | Treatment period: Day 8 (Pre-dose and 0-4, 4-8 and 8-12 hours post-dose)
  To assess Ae(t1-t2) after administration of multiple dose of AZD9977 oral suspension.
Urine PK parameter: Percentage Fraction of dose excreted in urine from time t1 to t2 (fe[t1-t2]%) | Treatment period: Day 8 (Pre-dose and 0-4, 4-8 and 8-12 hours post-dose)
  To assess fe(t1-t2)% after administration of multiple dose of AZD9977 oral suspension.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Harrow, United Kingdom

IPD SHARING:
Plan to Share IPD: No